CLINICAL TRIAL: NCT02896257
Title: De-implementing Inhaled Steroids to Improve Care and Safety in COPD (DISCUSS COPD) (QUE 15-471)
Brief Title: De-implementing Inhaled Steroids to Improve Care and Safety in COPD
Acronym: DISCUSS COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: QUX 16-009; QUE 15-271 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2016-08-12; First posted 2016-09-12 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Treatment of Chronic Obstructive Pulmonary Disease
Keywords: Quality Improvement; Quality Enhancement Research Initiatives; QuERI; Interventional; Multicenter; Inhaled corticosteroids; Pneumonia; Safety; De-implementation; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive; Pulmonary Diseases, Chronic Obstructive COPD
MeSH Terms: conditions — Pneumonia; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proactive patient-tailored electronic consult (E-consult) (Other): Primary care clinicians receive patient-tailored guideline concordant treatment recommendations, including orders and rationale to discontinue inhaled corticosteroids.
  Interventions: Other: Guideline treatment recommendations
- Usual care (No Intervention): Standard practice (usual care). Primary care providers treat their patients as usual.

INTERVENTIONS:
Other: Guideline treatment recommendations — Patient-tailored E-consult, orders and rationale to discontinue inhaled corticosteroids and discontinue or receive other COPD related care.
  Arms: Proactive patient-tailored electronic consult (E-consult)

SUMMARY:
This Quality Enhancement Research Initiative (QuERI) project is designed to determine efficacy and acceptance of an intervention method to provide primary care providers with patient-tailored electronic consults and corresponding unsigned orders for de-implementation of inhaled corticosteroids (ICS) for patients with COPD when ICS are not indicated by guidelines.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is among the most common medical diagnoses among Veterans. Approximately half of those who carry a diagnosis of COPD are prescribed inhaled corticosteroids (ICS), despite ICS having no role among those patients without fixed airflow obstruction (AFO) and a limited role among those who do. Guidelines explicitly state that ICS for COPD patients should be limited to those with severe AFO and those with frequent exacerbations. Even this benefit comes at a cost, as ICS use has been shown in multiple randomized controlled trials to increase rates of pneumonia. After prolonged exposure, ICS is also associated with higher bone fracture risk, incidence of cataracts and poor diabetes control. Among patients without disease or with mild-moderate AFO and low risk of exacerbation, ICS have no demonstrated efficacy, but retain the risk of harm. For this reason, evidence-based guidelines specifically recommend against their use in mild-moderate AFO.

The goal of this project is to improve the delivery and safety of care by de-implementing the ineffective use of ICS among Veterans with a diagnosis of COPD who otherwise lack a clinical indication for the medication. The primary aim is to reduce ICS use among Veterans with limited clinical indication for the medication. Investigators will test an intervention to de-implement unnecessary use of inhaled corticosteroids in Veterans with chronic obstructive pulmonary disease (COPD) by having pulmonologists assume more responsibility for supporting COPD patients. The investigators will compare a substitution approach using proactive patient-tailored electronic consult (E-consult) compared to usual care with a single-session education outreach, which represents a non-intensive unlearning approach. The investigators are targeting the intervention to Patient Aligned Care Team (PACT) providers who are randomized to either receive the intervention or not receive the intervention. For patients within intervention PACTs, the project clinicians will leverage the VA's integrated healthcare informatics system using specialist support through proactive patient-tailored electronic consults (E-consult) and inputting unsigned orders on behalf of Primary Care Providers (PCPs) to recommend and facilitate de-implementation of ICS. Primary care providers will have final say in accepting (signing), modifying, or declining the recommendations.

ELIGIBILITY:
Inclusion Criteria:

Provider:

Primary care provider (medical doctor/osteopathic physician, nurse practitioner, physician assistant [MD/DO, NP, PA]) assigned to a PACT from VA Puget Sound Health Care System or Edith Nourse Rogers Memorial Veterans Hospital (Bedford VA).

Patient:

* Patient is a Veteran who is assigned a VA PCP and has received Rx for an inhaled corticosteroid within the past 180 days.
* Patient has an inpatient or outpatient diagnosis of COPD in the prior two years.
* Patient has undergone spirometry in the past 5 years that indicates either no airflow obstruction or mild to moderate airflow obstruction indicated by a forced expiratory volume 1 (FEV1)/[greater of forced vital capacity (FVC) or vital capacity (VC)] =< 0.7 & FEV1% predicted >= 30%.

Exclusion Criteria:

Patients:

* Very severe airflow obstruction (<30% FEV1 % predicted)
* Severe disease as indicated by 1 inpatient COPD exacerbation in the year prior
* Severe disease as indicated by 2 outpatient COPD exacerbations in the year prior
* International Classification of Diseases (ICD) 9 and/or 10 diagnosed or clinically indicated asthmatics
* Significant bronchodilator response on spirometry (>12% increase in FEV1 post bronchodilator; >375 mL post-bronchodilator improvement)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-09-06 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Au, MD MS, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Christian D. Helfrich, PhD MPH BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to study start, we stratified all primary care teams based on site, provider type, and median number of eligible patients. Primary care teams were the unit of randomization, and providers were randomized along with their primary care team in a 1:1 ratio. For new providers, the unit of randomization was at the level of the PCP (stratified by site, provider type and median number of eligible patients).Only PCPs were considered enrolled. Patients were not considered enrolled in this study.
Pre-assignment Details: Prior to study start, we identified 139 primary care teams eligible for randomization; 2 primary care teams lost their associated provider prior to study start, leaving 137 primary care teams for initial randomization. Periodically, the Corporate Data Warehouse was queried to determine active primary care providers(PCPs) and their care teams. New PCPs and new care teams were added, resulting in a total of 220 distinct PCP-primary care team combinations.
Units Other Than Participants: PCP-Primary Care Teams
Groups:
- Usual Care: Primary care providers treat their patients as usual.
- Intervention: Primary care clinicians receive patient-tailored guideline concordant treatment recommendations, including orders and rationale to discontinue inhaled corticosteroids.
Period: Providers
Arm/Group | Usual Care | Intervention
Started | 88; 111 PCP-Primary Care Teams | 93; 109 PCP-Primary Care Teams
PCPs Assigned to 1 Primary Care Team | 68; 68 PCP-Primary Care Teams | 79; 79 PCP-Primary Care Teams
PCPs Assigned to Two Primary Care Teams | 18; 36 PCP-Primary Care Teams | 12; 24 PCP-Primary Care Teams
PCPs Assigned to 3 Primary Care Teams | 1; 3 PCP-Primary Care Teams | 2; 6 PCP-Primary Care Teams
PCPs Assigned to Four Primary Care Teams | 1; 4 PCP-Primary Care Teams | 0; 0 PCP-Primary Care Teams
Completed | 67; 76 PCP-Primary Care Teams | 65; 72 PCP-Primary Care Teams
Not Completed | 21; 35 PCP-Primary Care Teams | 28; 37 PCP-Primary Care Teams
Not completed — Without eligible patients | 21 | 28
Period: Patients
Arm/Group | Usual Care | Intervention
Started | 344; 111 PCP-Primary Care Teams (Eligible patient participants assigned to a usual care PCP=344) | 342; 109 PCP-Primary Care Teams (Eligible patient participants assigned to an intervention PCP=342)
Completed | 281; 76 PCP-Primary Care Teams (Patients with an eligible primary care appointment with a usual care PCP who were assigned an index date=281) | 269; 72 PCP-Primary Care Teams (Patients with an eligible primary care appointment with an intervention PCP who were assigned an index date=269)
Not Completed | 63; 35 PCP-Primary Care Teams | 73; 37 PCP-Primary Care Teams
Not completed — PFT entry criteria not met | 43 | 50
Not completed — No capacity to review | 8 | 11
Not completed — Appointment rescheduled/cancelled | 5 | 7
Not completed — PCP not assigned a clinic | 4 | 0
Not completed — No history of COPD | 0 | 1
Not completed — Deceased between review and index date | 0 | 1
Not completed — No ICS Rx upon review | 1 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Hospice care | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for age, sex, ethnicity, race not collected from primary care providers.
Groups:
- Usual Care Patients; Usual Care Providers: Standard practice (usual care). Primary care providers treat their patients as usual.
- Intervention Patients; Intervention Providers: Primary care clinicians receive patient-tailored guideline concordant treatment recommendations, including orders and rationale to discontinue inhaled corticosteroids.
  Guideline treatment recommendations: Patient-tailored E-consult, orders and rationale to discontinue inhaled corticosteroids and discontinue or receive other COPD related care.
- Total: Total of all reporting groups
Arm/Group | Usual Care Patients | Intervention Patients | Usual Care Providers | Intervention Providers | Total
Number analyzed (Participants) | 281 | 269 | 88 | 93 | 731
Age, Categorical [Count of Participants; unit: Participants] — Population: Data not collected from providers.
  Participants
    number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    <=18 years | 0 | 0 |  |  | 0
    Between 18 and 65 years | 75 | 58 |  |  | 133
    >=65 years | 206 | 211 |  |  | 417
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data not collected from providers.
  years
    number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    (all) | 69.1 (8.8) | 70.7 (9.0) |  |  | 69.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected from providers.
  Participants
    number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    Female | 7 | 5 |  |  | 12
    Male | 274 | 264 |  |  | 538
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected from providers.
  Participants
    number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    Hispanic or Latino | 4 | 5 |  |  | 9
    Not Hispanic or Latino | 271 | 257 |  |  | 528
    Unknown or Not Reported | 6 | 7 |  |  | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected from providers.
  Participants
    number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    American Indian or Alaska Native | 2 | 5 |  |  | 7
    Asian | 1 | 1 |  |  | 2
    Native Hawaiian or Other Pacific Islander | 4 | 1 |  |  | 5
    Black or African American | 15 | 12 |  |  | 27
    White | 244 | 227 |  |  | 471
    More than one race | 0 | 0 |  |  | 0
    Unknown or Not Reported | 15 | 23 |  |  | 38
Region of Enrollment [Count of Participants; unit: Participants] — Population: Data not collected from providers.
  Participants
    United States: number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    United States | 281 | 269 |  |  | 550
Smoking [Count of Participants; unit: Participants] — Population: Data not collected from providers.
  Participants
    number analyzed (Participants) | 281 | 269 | 0 | 0 | 550
    Former or Never Smoker | 155 | 162 |  |  | 317
    Current Smoker | 115 | 93 |  |  | 208
    Missing | 11 | 14 |  |  | 25
Provider type [Count of Participants; unit: Participants] — Population: Data not applicable to patient participants.
  Participants
    number analyzed (Participants) | 0 | 0 | 88 | 93 | 181
    Physicians |  |  | 57 | 60 | 117
    Advanced Practice Providers |  |  | 31 | 33 | 64
Site [Count of Participants; unit: Participants]
  Site 1 | 67 | 57 | 12 | 12 | 148
  Site 2 | 214 | 212 | 76 | 81 | 583
Mean number of eligible patients [Mean (Standard Deviation); unit: number of patients] — Mean number of potentially eligible patients assigned to the PCP at time of randomization. Population: Data not applicable to patient participants.
  number of patients
    number analyzed (Participants) | 0 | 0 | 88 | 93 | 181
    (all) |  |  | 4.0 (3.5) | 4.1 (3.6) | 4.1 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Discontinued or Expired and Not Renewed Inhaled Corticosteroids That Remain Off at 6 Months.
Description: Percentage of patients with discontinued or expired and not renewed inhaled corticosteroids that remain off at 6 months from index date.
Time Frame: Assessed at 6 months post primary care visit defined as (index date + 180 days)
Population: Patient participants that are assigned to usual care or intervention primary care providers.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 281 | 269
Participants | 94 | 174
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority; p < 0.001, Regression, Logistic; Mixed-random effects for provider clustering and adjusting for smoking status. Multiple imputation by chained equations for missing smoking status; Odds Ratio (OR) = 3.66, 95% CI 2-sided [2.50 to 5.38]

2. Secondary Outcome: Rate of COPD Exacerbation
Description: Rate of COPD exacerbation within 6 months starting the day after index date.
Time Frame: Within 6 months defined as (index date +1 day) to (index date + 180 days)
Population: Patient participants that are assigned to usual care or intervention primary care providers. One patient in the intervention group died between clinical review and the index date and was excluded from this analysis.
Measure: Number; unit: Events per 6 months of person-time
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 281 | 268
Events per 6 months of person-time | 0.11 | 0.09
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority; p = 0.47, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.44 to 1.47]

3. Secondary Outcome: Rate of Pneumonia
Description: Rate of pneumonia within 6 months starting the day after index date.
Time Frame: Within 6 months defined as (index date +1 day) to (index date + 180 days)
Population: as for outcome 2
Measure: Number; unit: Events per 6 months of person-time
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 281 | 268
Events per 6 months of person-time | 0.03 | 0.02
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority; p = 0.42, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.20 to 1.96]

4. Secondary Outcome: Mortality
Description: Mortality determined by the presence of date of death occurring between (index date + 1 day) to (index date + 180 days)
Time Frame: Assessed during 6 months following primary care visit defined as (index date + 1 day) to (index date + 180 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 281 | 268
Participants | 9 | 10

5. Secondary Outcome: Number of Patients Recommended to Stop Inhaled Corticosteroids
Description: Among patients of intervention PCPs, number of patients recommended to stop inhaled corticosteroids
Time Frame: Collected at time of recommendation/order entry
Population: Patient participants assigned to intervention PCPs.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 269
Participants | 181

6. Secondary Outcome: Percentage of Recommendations to Discontinue Inhaled Corticosteroids Accepted by Primary Care Providers
Description: Among patients assigned to intervention PCPs, percentage of recommendations to discontinue inhaled corticosteroids accepted by primary care providers
Time Frame: Assessed during 6 months following index date
Population: Recommendations to discontinue inhaled corticosteroids. A recommendation to discontinue inhaled corticosteroids was made only once per patient.
Measure: Number; unit: Percentage of recommendations
Arm/Group | Intervention
Number analyzed (Participants) | 181
Percentage of recommendations | 92.3

7. Secondary Outcome: Percentage of Patients Where ICS Discontinuation Recommendations Are Accepted But Restarted by 6 Months Following Index Date
Description: Percentage of patients where ICS discontinuation recommendations are accepted but restarted by 6 months following index date
Time Frame: Assessed at 6 months post index date
Population: Patients where ICS discontinuation recommendation was accepted.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 167
Participants | 24

8. Secondary Outcome: Number of Patients for Whom Recommendations Are Made
Description: Among patients assigned to intervention providers, number of patients for whom recommendations are made.
Time Frame: Collected at time or recommendation order entry
Population: We identified 269 patients meeting entry and exclusion criteria cared for by a primary care provider assigned to the intervention group. Of these, 262 received an electronic consult with recommendations for guideline concordant COPD care.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 269
Participants | 262

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not collected from providers.
Groups:
- Intervention: Primary care clinicians receive patient-tailored guideline concordant treatment recommendations, including orders and rationale to discontinue inhaled corticosteroids.
  Guideline treatment recommendations: Patient-tailored E-consult, orders and rationale to discontinue inhaled corticosteroids and discontinue or receive other COPD related care.
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 9/281 | 10/269
Serious Adverse Events (participants affected / at risk) | 41/281 | 30/269
Other Adverse Events (participants affected / at risk) | 0/281 | 0/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=281) | Intervention (N=269)
Inpatient COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 6 | 7 — Hospitalized for COPD exacerbation within the 180 days after the index date.
Outpatient COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 30 | 23 — Experienced an outpatient COPD exacerbation within the 180 days after the index date.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 | 5 — Experienced either an inpatient or outpatient pneumonia event within 180 days after the index date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02896257/Prot_SAP_000.pdf